CLINICAL TRIAL: NCT02663973
Title: Prospective Evaluation of Breast Cancer at Brazilian Institutions - Project AMAZONA III
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Avon Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: GBECAM 0115
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The principal goal of this study is to describe the epidemiology of breast cancer in the Brazilian population

DETAILED DESCRIPTION:
The principal goal of this study is to describe the epidemiology of breast cancer in the Brazilian population. Other specific goals are:

* To evaluate the demographic and socio-demographic profile, comorbidities and reproductive risks, anthropometric profile and family history.
* Characterize the breast tumors immunophenotype through anatomopathological data, such as: tumor grade, estrogen receptor, progesterone receptor, HER2, Ki67.
* Describe the screening tests, main symptoms and cancer stage in the moment of the diagnosis.
* Describe the initial cancer treatment and locally advanced such as surgery, radiotherapy, chemotherapy and endocrine therapy.
* Describe palliative treatment for recurrent or metastatic breast cancer: chemotherapy, radiotherapy, biphosphonate, and others.
* Evaluate the clinical outcomes such as: local or diffuse relapse, period of time until progression to metastatic cancer, global lifespan and specific breast cancer lifespan.
* Evaluate clinical complications of the metastatic disease, such as: brain metastasis, spinal cord compression, skeletal related events.
* Analyze the demographical and socio-economical characteristics, clinical-pathological characteristics of the tumor, treatment, clinical outcomes, type of institution (private/public), and other factors that may impact clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 18 years old
* Invasive breast cancer stage I to IV proven by histology or cytology
* Patients with new pathological diagnosis of invasive primary BC after the site activation date
* Pathological diagnosis of invasive breast cancer during recruitment (6 months before center activation or until 3000 patients included)
* New primary cancer on the same breast or contralateral breast.
* Patient's medical chart is available and adequate for data collection
* Patient properly signed the informed consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Woman ≥ 18 years old with recent diagnosis of breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2016-01-01; Primary Completion 2020-06-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Description of the epidemiology of breast cancer in the Brazilian population | Annually, during 5 years

SECONDARY OUTCOMES:
Description of the socioeconomical characteristics of the Brazilian population with breast cancer | Annually, during 5 years
Characterization of the immunophenotypic markers of the tumor | Annually, during 5 years
  estrogen receptor, progesterone receptor, HER2, Ki67
Classification of breast cancer staging | Annually, during 5 years
Description of screening tests of breast cancer patients in Brazil | Annually, during 5 years
Main symptoms presented by patients with breast cancer in Brazil | Annually, during 5 years
Initial treatment for breast cancer of Brazilian patients | Annually, during 5 years
Type of palliative treatment for metastasis or recurrent breast cancer in Brazilian patients | Annually, during 5 years
Clinical outcome of Brazilian breast cancer patients | Annually, during 5 years
Types of clinical complications displayed by breast cancer Brazilian patients | Annually, during 5 years
Characterization of exterior factors that may impact clinical outcome of breast cancer Brazilian patients | Annually, during 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Werutsky, MD, Study Director — Latin American Cooperative Oncology Group
Locations (24):
- Brazil (24):
  - Centro Regional Integrado de Oncologia (CRIO), Fortaleza, Ceará
  - Clínica AMO, Salvador, Estado de Bahia
  - Núcleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Centro de Pesquisa do Setor de Ginecologia e Mama do Hospital Araújo Jorge, Goiânia, Goiás
  - Unidade de Pesquisa Clínica/Hospital de Clínicas da UFG, Goiânia, Goiás
  - Unidade de Pesquisa Clínica do Hospital do Câncer de Londrina, Londrina, Paraná
  - Hospital Jardim Amália, Volta Redonda, Rio de Janeiro
  - Centro de Pesquisa Clínica da Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - Centro de Pesquisas da Serra Gaúcha, Caxias do Sul, Rio Grande do Sul
  - Instituto de Pesquisa Clínicas para Estudos Multicêntricos da UCS, Caxias do Sul, Rio Grande do Sul
  - Hospital da Cidade de Passo Fundo - Clínica CITO, Passo Fundo, Rio Grande do Sul
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Grupo de Estudos em Pesquisa de Pelotas, Pelotas, Rio Grande do Sul
  - CPO - Pucrs, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Novos Tratamentos em Câncer - Hospital Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - CEPON, Florianópolis, Santa Catarina
  - Clínica de Neoplasias Litoral - Centro de Novos Tratamentos Itajaí, Itajaí, Santa Catarina
  - Instituto Oncológico de Ribeirão Preto - InORP, Ribeirão Preto, São Paulo
  - Instituto Nacional do Câncer, Rio de Janeiro
  - Oncoclínica, Rio de Janeiro
  - Centro de Pesquisa Clínica do Hospital Israelita Albert Einstein, São Paulo
  - Centro de Pesquisa Instituto do Câncer Arnaldo Vieira de Carvalho, São Paulo
  - Hospital AC Camargo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allemani C, Weir HK, Carreira H, Harewood R, Spika D, Wang XS, Bannon F, Ahn JV, Johnson CJ, Bonaventure A, Marcos-Gragera R, Stiller C, Azevedo e Silva G, Chen WQ, Ogunbiyi OJ, Rachet B, Soeberg MJ, You H, Matsuda T, Bielska-Lasota M, Storm H, Tucker TC, Coleman MP; CONCORD Working Group. Global surveillance of cancer survival 1995-2009: analysis of individual data for 25,676,887 patients from 279 population-based registries in 67 countries (CONCORD-2). Lancet. 2015 Mar 14;385(9972):977-1010. doi: 10.1016/S0140-6736(14)62038-9. Epub 2014 Nov 26. PMID 25467588
- [Background] Freitas-Junior R, Gonzaga CM, Freitas NM, Martins E, Dardes Rde C. Disparities in female breast cancer mortality rates in Brazil between 1980 and 2009. Clinics (Sao Paulo). 2012 Jul;67(7):731-7. doi: 10.6061/clinics/2012(07)05. PMID 22892915
- [Background] Gonzaga CM, Freitas-Junior R, Souza MR, Curado MP, Freitas NM. Disparities in female breast cancer mortality rates between urban centers and rural areas of Brazil: ecological time-series study. Breast. 2014 Apr;23(2):180-7. doi: 10.1016/j.breast.2014.01.006. Epub 2014 Feb 4. PMID 24503143
- [Background] Palmer JR, Viscidi E, Troester MA, Hong CC, Schedin P, Bethea TN, Bandera EV, Borges V, McKinnon C, Haiman CA, Lunetta K, Kolonel LN, Rosenberg L, Olshan AF, Ambrosone CB. Parity, lactation, and breast cancer subtypes in African American women: results from the AMBER Consortium. J Natl Cancer Inst. 2014 Sep 15;106(10):dju237. doi: 10.1093/jnci/dju237. Print 2014 Oct. PMID 25224496
- [Background] Phipps AI, Chlebowski RT, Prentice R, McTiernan A, Wactawski-Wende J, Kuller LH, Adams-Campbell LL, Lane D, Stefanick ML, Vitolins M, Kabat GC, Rohan TE, Li CI. Reproductive history and oral contraceptive use in relation to risk of triple-negative breast cancer. J Natl Cancer Inst. 2011 Mar 16;103(6):470-7. doi: 10.1093/jnci/djr030. Epub 2011 Feb 23. PMID 21346227
- [Background] Anderson KN, Schwab RB, Martinez ME. Reproductive risk factors and breast cancer subtypes: a review of the literature. Breast Cancer Res Treat. 2014 Feb;144(1):1-10. doi: 10.1007/s10549-014-2852-7. Epub 2014 Jan 30. PMID 24477977
- [Background] Vona-Davis L, Howard-McNatt M, Rose DP. Adiposity, type 2 diabetes and the metabolic syndrome in breast cancer. Obes Rev. 2007 Sep;8(5):395-408. doi: 10.1111/j.1467-789X.2007.00396.x. PMID 17716297
- [Background] Calle EE, Rodriguez C, Walker-Thurmond K, Thun MJ. Overweight, obesity, and mortality from cancer in a prospectively studied cohort of U.S. adults. N Engl J Med. 2003 Apr 24;348(17):1625-38. doi: 10.1056/NEJMoa021423. PMID 12711737
- [Background] Reeves GK, Pirie K, Beral V, Green J, Spencer E, Bull D; Million Women Study Collaboration. Cancer incidence and mortality in relation to body mass index in the Million Women Study: cohort study. BMJ. 2007 Dec 1;335(7630):1134. doi: 10.1136/bmj.39367.495995.AE. Epub 2007 Nov 6. PMID 17986716
- [Background] Cleveland RJ, Eng SM, Abrahamson PE, Britton JA, Teitelbaum SL, Neugut AI, Gammon MD. Weight gain prior to diagnosis and survival from breast cancer. Cancer Epidemiol Biomarkers Prev. 2007 Sep;16(9):1803-11. doi: 10.1158/1055-9965.EPI-06-0889. PMID 17855698
- [Background] Anders CK, Deal AM, Miller CR, Khorram C, Meng H, Burrows E, Livasy C, Fritchie K, Ewend MG, Perou CM, Carey LA. The prognostic contribution of clinical breast cancer subtype, age, and race among patients with breast cancer brain metastases. Cancer. 2011 Apr 15;117(8):1602-11. doi: 10.1002/cncr.25746. Epub 2010 Nov 29. PMID 21472708
- [Background] Perou CM, Sorlie T, Eisen MB, van de Rijn M, Jeffrey SS, Rees CA, Pollack JR, Ross DT, Johnsen H, Akslen LA, Fluge O, Pergamenschikov A, Williams C, Zhu SX, Lonning PE, Borresen-Dale AL, Brown PO, Botstein D. Molecular portraits of human breast tumours. Nature. 2000 Aug 17;406(6797):747-52. doi: 10.1038/35021093. PMID 10963602
- [Background] Liedke PE, Finkelstein DM, Szymonifka J, Barrios CH, Chavarri-Guerra Y, Bines J, Vasconcelos C, Simon SD, Goss PE. Outcomes of breast cancer in Brazil related to health care coverage: a retrospective cohort study. Cancer Epidemiol Biomarkers Prev. 2014 Jan;23(1):126-33. doi: 10.1158/1055-9965.EPI-13-0693. Epub 2013 Oct 28. PMID 24165578
- [Background] Lohman TG, Roche AF, Martorell R. Anthropometric standardization reference manual. Illinois: A division of human Kinetics Publishers Inc, 1988.
- [Derived] Werutsky G, Lopes M, de Jesus RG, Gazola AA, Pellegrini RA, Rebelatto TF, Freitas LVW, Heck AP, da Silva AF, Rodrigues MF, Gossling G, Giacomazzi J, Rocha MS, Rosa DD, Barrios CH, Cronemberger EH, Queiroz GS, Bines J, Simon SD, Fay AP. The impact of a breast cancer diagnosis on marital outcomes and factors associated with divorce and separation. Rev Bras Ginecol Obstet. 2024 Jun 27;46:e-rbgo60. doi: 10.61622/rbgo/2024rbgo60. eCollection 2024. PMID 38994465
- [Derived] Maschmann RM, De Jesus RG, Werutsky G, Rebelatto TF, Queiroz G, Simon SD, Bines J, Barrios CHE, Rosa DD. Time interval between diagnosis to treatment of breast cancer and the impact of health insurance coverage: a sub analysis of the AMAZONA III Study (GBECAM 0115). Breast Cancer Res Treat. 2023 Feb;198(1):123-130. doi: 10.1007/s10549-022-06809-8. Epub 2022 Dec 31. PMID 36586038
- [Derived] Franzoi MA, Rosa DD, Zaffaroni F, Werutsky G, Simon S, Bines J, Barrios C, Cronemberger E, Queiroz GS, Cordeiro de Lima V, Junior RF, Couto J, Emerenciano K, Resende H, Crocamo S, Reinert T, Van Eyli B, Neron Y, Dybal V, Lazaretti N, de Cassia Costamillan R, Pinto de Andrade DA, Mathias C, Vacaro GZ, Borges G, Morelle A, Filho CAS, Mano M, Liedke PER. Advanced Stage at Diagnosis and Worse Clinicopathologic Features in Young Women with Breast Cancer in Brazil: A Subanalysis of the AMAZONA III Study (GBECAM 0115). J Glob Oncol. 2019 Nov;5:1-10. doi: 10.1200/JGO.19.00263. PMID 31730380
- See also: World Health Organization. GLOBOCAN 2012: cancer incidence and mortality worldwide. Accessed in Jan 8 2015. — http://globocan.iarc.fr/Pages/fact_sheets_population.aspx
- See also: National Cancer Institute. Cancer treatment. Accessed in Jan 8 2015. — http://www.cancer.gov/cancertopics/treatment